CLINICAL TRIAL: NCT01282632
Title: A Double Blind Pilot Trial to Evaluate Efficacy Trends and Safety of Risperidone and Olanzapine as add-on Therapy to Serotonin Type Antidepressants in Subjects With Treatment Resistant Depression (TRD)
Brief Title: Risperidone vs. Olanzapine as add-on Treatment in Treatment Resistant Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Dr. Anthony Levitt, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ro123
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-09

CONDITIONS: Subjects Had Unipolar, Non-psychotic Major Depression
Keywords: depression; treatment resistant depression; unipolar; non- psychotic major depression; add-on to a serotonin type antidepressants; risperidone; olanzapine; double blind comparison; randomized
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant | interventions — Risperidone; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperidone (Experimental): Commence at 0.5 mg once daily Increase, blindly, to 1 mg and then by 1 mg at discretion of clinicians through weeks 1-4 to a maximum of 3 mg.
  Interventions: Drug: Risperidone
- Olanzapine (Experimental): Commence at 2.5 mg once daily Increase to 5.0 mg, blindly, and then by 5 mg at the discretion of the clinician through weeks 1 - 4 to a maximum of 15 mg
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Risperidone — Risperidone will commence at 0.5 mg per day in a single daily dose given once in the evening. Clinicians will have the option, at each visit of increasing the risperidone dose to a maximum of 3 mg/day based on subject response and tolerability (please see Titration Recommendations below).
  Arms: Risperidone
Drug: Olanzapine — Olanzapine will commence at 2.5 mg per day in a single daily dose given once in the evening. Clinicians will have the option, at each visit, of increasing the olanzapine dose to a maximum of 15 mg/day based on subject response and tolerability.
  Arms: Olanzapine

SUMMARY:
Atypical neuroleptics may have antidepressant qualities in bipolar depression and in unipolar depression. Some data support the use of both Risperidone and Olanzapine, but there are no direct comparisons of their relative efficacy and tolerability in treatment resistant depression. The current study was designed as a pilot study to examine efficacy and tolerability of Olanzapine vs. Risperidone add on to a failed serotonin re-uptake inhibitor (SSRI) in depression.

DETAILED DESCRIPTION:
Overview of Study Design

This is a Canadian, multicentre, double blind, comparator trial in 42 patients with TRD. TRD is defined as the failure to respond adequately to two successive courses of different antidepressants at an adequate dose (at least fluoxetine 20 mg, citalopram 20 mg, paroxetine 20 mg, sertraline 100 mg, fluvoxamine 150 mg, venlafaxine 225 mg)) for at least 4 weeks. All subjects, at entry to the study will be currently not responding to treatment of at least 4 weeks duration of a serotonin re-uptake inhibitor (SSRI) or a selective nor-epinephrine and serotonin re-uptake inhibitor (SNRI). Non-response is defined as a score of 3 ("minimal improvement") or worse on the Clinical global Impression of Improvement .

The objective is to assess the appropriateness of the trial design and to determine sample size requirements for future controlled trials. In addition the efficacy and safety of oral doses of risperidone (.5-3 mg/day) and olanzapine (2.5-15 mg.day) as add-on therapy to any SSRI or SNRI in treatment resistant depression will be evaluated. Subjects meeting the screening criteria will enter a 6-week trial with risperidone or olanzapine added on to the current SSRI or SNRI therapy.

A medical/ psychiatric history, HAM-D-29 (only the first 17 items will be used for outcome), MADRS and HAM-A will be obtained at screening. At subsequent visits HAM-D, HAM-A, and MADRS will be performed and adverse events (spontaneous and using the CASES checklist) and concomitant medications will be collected.

Recruitment:

Subjects will drawn from two sources:

1. Outpatients currently attending the clinic at the sites. These subjects will already be in treatment or may have been referred from the local communities of the clinics involved in this study for consultation. Should these subjects drop out or once they have completed the study they will receive the treatment as usual at each site.
2. Advertisements. Advertisements will be placed in local media (radio, television, newspaper) identifying the nature of the study and providing a contact number. These advertisements will be approved by the local IRB's prior to posting.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are eligible for this trial:

1. Male or female out-patients;
2. Aged between 18 and 65 years (extremes included);
3. Subjects suffering from a current episode of non-psychotic, unipolar depression as determined by the depression section of the SCID-IV.
4. Subjects with treatment resistant depression defined as failure to respond to two successive courses of monotherapy given in adequate doses for a minimum of 4 weeks with different antidepressants (the current course of antidepressant can be considered to second failed course) and;
5. Subjects currently taking a SSRI or a SNRI for at least 4 weeks, at adequate dosage and not responding, as defined by a score of 3 or more on the CGI-I. and no dose change for 2 weeks prior to entry.
6. A minimum score of 16 on the 17 item HAM-D
7. Ability to provide informed consent.

Exclusion Criteria:

Subjects meeting one or more of the following criteria cannot be selected:

1. Subjects who are actively suicidal as determined by a score of 3 on the suicide item on the HAM-D or in the opinion of the treating physician;
2. Other current (active symptomatology within the last 2 months) Axis I DSM IV diagnosis other than nicotine or caffeine dependence or other than an Anxiety disorder.
3. Use of disallowed concomitant therapy; or other psychotropic medication except occasional benzodiazepines. (See "Rescue Medication");
4. History of alcohol or drug abuse or dependence, within 3 months of entry into the trial);
5. Seizure disorder requiring medication;
6. Active medical condition that requires urgent attention or that would contra-indicate the use of risperidone or olanzapine. For example stable thyroid disease or asthma would be acceptable, whereas acute hepatitis would not;
7. Participation in an investigational drug trial within 30 days prior to the start of the trial
8. Known sensitivity to risperidone, olanzapine or the antidepressant;
9. History of neuroleptic malignant syndrome (NMS);
10. Subjects who are at imminent risk of injury to self or others, or causing significant damage to property, as judged by the investigator;
11. Female subjects who are pregnant or breast-feeding;
12. Female subject of childbearing potential without adequate contraception (sterilization, barrier, IUD, oral contraceptives, intramuscular or subdermal administration of depot-progestagens);

15. Previous exposure to risperidone or olanzapine during the current episode.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-08; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hamilton Depression Rating Scale at 1 week | day one
  Subject to be eligible for this trial must have a minimum score of 16 on the 17 item HAM-D which will be obtained at screening. Efficacy will be measured on the HAM-D 17 and defined as a 50% decrease from baseline to week 6.
Change from Baseline in Montgomery Asberg Depression Scale (MADRS)at 1 week | day one
  MADRS will be obtained at screening. Efficacy will be measured by the MADRS and defined as a 50% decrease from baseline to week 6.
Change from baseline Hamilton Rating Scale for Anxiety (HAM-A) at 1 week | day one
  Impact on anxiety will be measured by the HAM-A over the 6 weeks.
Change from Baseline in Hamilton Depression Rating Scale at 2 weeks | day 8
  Subject to be eligible for this trial must have a minimum score of 16 on the 17 item HAM-D which will be obtained at screening. Efficacy will be measured on the HAM-D 17 and defined as a 50% decrease from baseline to week 6.
Change from Baseline in Hamilton Depression Rating Scale at 3 weeks | day 15
  Subject to be eligible for this trial must have a minimum score of 16 on the 17 item HAM-D which will be obtained at screening. Efficacy will be measured on the HAM-D 17 and defined as a 50% decrease from baseline to week 6.
Change from Baseline in Hamilton Depression Rating Scale at 4 weeks | day 22
  Subject to be eligible for this trial must have a minimum score of 16 on the 17 item HAM-D which will be obtained at screening. Efficacy will be measured on the HAM-D 17 and defined as a 50% decrease from baseline to week 6.
Change from Baseline in Hamilton Depression Rating Scale at 5 weeks | day 29
  Subject to be eligible for this trial must have a minimum score of 16 on the 17 item HAM-D which will be obtained at screening. Efficacy will be measured on the HAM-D 17 and defined as a 50% decrease from baseline to week 6.
Change from Baseline in Hamilton Depression Rating Scale at 6 weeks | day 43
  Subject to be eligible for this trial must have a minimum score of 16 on the 17 item HAM-D which will be obtained at screening. Efficacy will be measured on the HAM-D 17 and defined as a 50% decrease from baseline to week 6.
Change from Baseline in Montgomery Asberg Depression Scale (MADRS)at 2 weeks | day 8
  MADRS will be obtained at screening. Efficacy will be measured by the MADRS and defined as a 50% decrease from baseline to week 6.
Change from Baseline in Montgomery Asberg Depression Scale (MADRS)at 3 weeks | day 15
  MADRS will be obtained at screening. Efficacy will be measured by the MADRS and defined as a 50% decrease from baseline to week 6.
Change from Baseline in Montgomery Asberg Depression Scale (MADRS)at 4 weeks | day 22
  MADRS will be obtained at screening. Efficacy will be measured by the MADRS and defined as a 50% decrease from baseline to week 6.
Change from Baseline in Montgomery Asberg Depression Scale (MADRS)at 5 weeks | day 29
  MADRS will be obtained at screening. Efficacy will be measured by the MADRS and defined as a 50% decrease from baseline to week 6.
Change from Baseline in Montgomery Asberg Depression Scale (MADRS)at 6 weeks | day 43
  MADRS will be obtained at screening. Efficacy will be measured by the MADRS and defined as a 50% decrease from baseline to week 6.
Change from baseline Hamilton Rating Scale for Anxiety (HAM-A) at 2 weeks | day 8
  Impact on anxiety will be measured by the HAM-A over the 6 weeks.
Change from baseline Hamilton Rating Scale for Anxiety (HAM-A) at 3 weeks | day 15
  Impact on anxiety will be measured by the HAM-A over the 6 weeks.
Change from baseline Hamilton Rating Scale for Anxiety (HAM-A) at 4 weeks | day 15
  Impact on anxiety will be measured by the HAM-A over the 6 weeks.
Change from baseline Hamilton Rating Scale for Anxiety (HAM-A) at 5 weeks | day 22
  Impact on anxiety will be measured by the HAM-A over the 6 weeks.
Change from baseline Hamilton Rating Scale for Anxiety (HAM-A) at 6 weeks | day 43
  Impact on anxiety will be measured by the HAM-A over the 6 weeks.

SECONDARY OUTCOMES:
Clinical Global Improvement Scale - Improvement | day one
  Subjects currently taking a SSRI or a SNRI for at least 4 weeks, at adequate dosage and not responding, as defined by a score of 3 or more on the CGI-I.
Change from Baseline of Weight at 6 weeks | day 43
  Weight (Kg) will be measured with subjects at screening then at week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Levitt, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Raymond Lam, MD, Study Director — University of British Columbia; Yves Chaput, MD, Study Director — University of Manitoba; Murray Enns, MD, Study Director — University of McGill
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada